CLINICAL TRIAL: NCT02934516
Title: Delivery of Impacted Fetal Head During Cesarean Section for Obstructed Labor: Push Method Versus Abdominal Disimpaction With Lower Uterine Segment Support
Brief Title: Push With Lower Uterine Segment Support
Acronym: PLUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Aswan University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, M.B.B.Ch, M.Sc, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLUS-DIH-02
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Dystocia
Keywords: Obstructed labor; C section. push method; reverse breech
MeSH Terms: conditions — Dystocia | interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disimpaction with lower uterine support (Experimental): Cesarean section with support of the lower uterine segment
  Interventions: Procedure: Cesarean section
- Classic push method (Active Comparator): Cesarean section with push method
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — Abdominal disimpaction with lower uterine segment support: the edge of the lower uterine segment is grasped by 3-4 modified Allies forceps (with broader jaws) applied along the lower edge of the incision until it is completely supported. These forceps are handled by the assistant, and gentle traction is applied upward, perpendicular to the uterine surface and away from the fetal head without excessive force. Accordingly, the hand of the surgeon could be inserted into the uterine cavity, and adequate space for manipulations is available without applying pressure on the lower segment. The fetal head is eventually grasped and delivered.
  Classic push method: delivering the head with assistance by pushing the fetal head vaginally

SUMMARY:
The study aims to compare maternal and early neonatal outcomes of abdominal disimpaction with lower uterine segment support in comparison to the classic "push" method for delivery of impacted fetal head during Cesarean section for obstructed labor.

DETAILED DESCRIPTION:
Obstructed labor refers to failure of labor progress in spite of good uterine contractions and is attributed to mismatch between the size of the presenting part of the fetus and the mother's pelvis. Approximately 8% of maternal deaths worldwide are attributed to obstructed labor and subsequent puerperal infection, uterine rupture, and postpartum hemorrhage.

In these situations, Cesarean section could minimize maternal and neonatal morbidity. However, Cesarean section is challenging when the head is deeply impacted and is associated with high risk of maternal injuries and perinatal injuries. The most common complication is extension of uterine incision which could involve the vagina, bladder, ureters and broad ligament. Neonates are also at risk of skull fractures, cephalhematoma, and subgaleal hematoma mainly due to manipulations. Currently, the most popular approaches for fetal head delivery are the push and pull methods. Although push method seems to be more convenient and does not necessitate extensive experience, it is more significantly associated with extension than the pull method. Although pull method seems to be more safe, it is more difficult to perform and usually warrants an aggressive uterine incision to deliver the fetus. In 2013, investigators published a case series on abdominal disimpaction with lower uterine segment support which basically allows obstetricians to deliver the fetal head through a transverse uterine incision with minimal risk of extensions and neonatal complications. In this study, investigators aim to validate this approach in comparison to the classic push method.

ELIGIBILITY:
Inclusion Criteria:

* Singleton term pregnancy, 37 to 42 weeks of gestation.
* Cephalic presentation.
* The cervix is fully dilated.
* Ruptured membranes.
* Adequate uterine contractions.
* Impacted fetal head in maternal pelvis

Exclusion Criteria:

* Intrauterine fetal death
* Major fetal anomalies
* Non-cephalic presentation
* Multiple pregnancy
* Preterm caesarean < 37 weeks
* Abnormal placentation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Extension of uterine incision | During delivery of the fetus
  The incidence of extension of uterine incision
Length of extension of uterine incision | During delivery of the fetus
  If extension of uterine incision happens, the length of extension will be measured
Injury of the vagina | During delivery of the fetus
  Extension of uterine incision into the vagina
Injury of the bladder | During delivery of the fetus
  Extension of uterine incision into the bladder
Injury of the ureter | During delivery of the fetus
  Extension of uterine incision into the ureter

SECONDARY OUTCOMES:
Cesarean section operative time | Time from incision to closure of the skin (within 24 hours of recruitment)
  Duration of Cesarean section operation
Intra-operative blood loss | During Cesarean section only
  Amount of blood loss as estimated by suction device from incision to closure of the skin
The incidence of postpartum hemorrhage | During the first 24 hours post-operative
  Loss of more than 500 ml during the first 24 hours after surgery and the management that will be done
Incidence of blood transfusion | During surgery and within the first 24 hours postoperative
  The incidence of blood transfusion due to significant blood loss (based on blood loss and clinical judgement "hypotension, tachycardia, pallor")
Fetal traumatic birth injuries | During Cesarean section (fetal delivery)
  Skull fractures, limb fractures, brachial plexus injury, cephalhematoma, and subgaleal hematoma
APGAR score | At 1 and 5 minutes after delivery of the newborn
Need for neonatal admission to neonatal intensive care unit | Within 24 hours of delivery of the newborn
Postoperative infections | 1 week of postpartum
  Puerperal sepsis and Cesarean section wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nasr, MBBCh, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolea C, AbouZahr C. Global burden of obstructed labour in the year 2000. World Health Organization (WHO), Geneva, Switzerland. 2003 Jul;1:17.
- [Background] Neilson JP, Lavender T, Quenby S, Wray S. Obstructed labour. Br Med Bull. 2003;67:191-204. doi: 10.1093/bmb/ldg018. PMID 14711764
- [Background] Landesman R, Graber EA. Abdominovaginal delivery: modification of the cesarean section operation to facilitate delivery of the impacted head. Am J Obstet Gynecol. 1984 Mar 15;148(6):707-10. doi: 10.1016/0002-9378(84)90551-9. PMID 6702937
- [Background] Shazly SA, Elsayed AH, Badran SM, Abdel Badee AY, Ali MK. Abdominal disimpaction with lower uterine segment support as a novel technique to minimize fetal and maternal morbidities during cesarean section for obstructed labor: a case series. Am J Perinatol. 2013 Sep;30(8):695-8. doi: 10.1055/s-0032-1331031. Epub 2012 Dec 27. PMID 23271386